CLINICAL TRIAL: NCT03828383
Title: Developing and Evaluating In-Home Supportive Technology for Dementia Caregivers
Brief Title: In-Home Technology for Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other); People Power Company (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert Levenson, Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R44AG059458 (NIH); R44AG059458 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Dementia; Alzheimer's Disease; Frontotemporal Dementia
Keywords: Caregivers; Dementia; In-Home Assistive Technology
MeSH Terms: conditions — Dementia; Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Identical system is installed in all homes regardless of treatment arm. The member of research team who does the installation will now know which treatment arm has been assigned. Initiating the features of the system appropriate to the assigned treatment arm is done remotely by a member of the People Power staff (who has no contact with the participants) following the installation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Home Technology System (Experimental): The full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) will be installed in the homes of caregivers by a member of the research team (blind as to arm of the study). Monitoring of sensors, provision of warnings, messaging, and social networking features will be activated remotely for those participants who have been randomly assigned to this arm. Participation will extend over a nine month period with questionnaires (e.g., health and well-being) administered 4 times (at the time of installation and every 3 months thereafter).
  Interventions: Device: In-home technology
- Limited In-Home Technology System (Sham Comparator): The full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) will be installed in the homes of caregivers by a member of the research team (blind as to arm of the study). Monitoring of the water leak sensor and associated warnings will be activated remotely for those participants who have been randomly assigned to this arm. Participation will extend over a nine month period with questionnaires (e.g., health and well-being) administered 4 times (at the time of installation and every 3 months thereafter).
  Interventions: Device: Limited in-home technology

INTERVENTIONS:
Device: In-home technology — Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using a trusted circle of friends and family who are encouraged to stay in contact and share photos and videos with the caregiver and person with dementia via the digital display.
  Arms: In-Home Technology System
Device: Limited in-home technology — Intelligent bot monitors the in-home water leak sensor and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome conditions occur.
  Arms: Limited In-Home Technology System

SUMMARY:
This study aims to develop and evaluate in-home assistive technology that is designed to alleviate anxiety, burden, and loneliness in spousal and familial caregivers of individuals with Alzheimer's disease and frontotemporal dementia.

DETAILED DESCRIPTION:
This study aims to develop, refine, and evaluate a hardware/software system designed to integrate in-home sensors and devices, social connection, and Internet-of-Things (i.e., devices that can be controlled and communicated with via the internet) technologies to create a more supportive and safe home environment for caregivers and people with dementia. The system monitors troublesome behaviors in people with dementia (e.g., wandering), and targets mechanisms (e.g., worry, social isolation) thought to link behavioral symptoms in people with dementia with adverse caregiver outcomes (declines in health and well-being). The system is designed to minimize demands on caregivers' limited time and energy and to provide a platform for data collection that can be used by researchers and care professionals.

Hypotheses:

1. Caregivers in the full operation condition will have fewer negative effects of caregiving (lower burden, higher mental and physical health, higher well-being) than those in the limited home safety condition.
2. Greater use of the social networking features of the system will be associated with fewer caregiver depressive symptoms.
3. Greater utilization of the home safety features of the system will be associated with fewer caregiver anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers are fluent/literate in English
* Caregivers currently reside with spouse/family member with dementia
* Caregivers primarily use an iPhone
* Caregiver has wireless internet in home

Exclusion Criteria:

* Caregivers providing care for individuals with known non-neurodegenerative conditions affecting behavior and cognition
* Caregivers providing care for individuals with longstanding Axis I psychiatric disorder
* Caregivers providing care for individuals with metabolic disorder or major organ dysfunction
* Caregivers providing care for individuals with alcohol abuse or dependence (within 5 years of dementia onset)
* Caregivers providing care for individuals with head trauma with loss of consciousness greater than 30 minutes
* Caregivers providing care for individuals with contraindications to MRI imaging
* Caregivers providing care for individuals with large confluent white matter lesions
* Caregivers providing care for individuals with significant systemic medical illness
* Caregivers providing care for individuals who use a medication likely to affect central nervous system functions adversely

If you live in the San Francisco Bay Area, Las Vegas (Clark County), Orange County, Los Angeles County, or Oregon, you may complete the following screening questionnaire to determine your eligibility for participation: https://bit.ly/UCBDC Upon completion of the screening questionnaire, the UC Berkeley research team will follow up soon after by email or phone to confirm your eligibility status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Levenson, Ph.D., Study Director — University of California, Berkeley
Locations (5):
- United States (5):
  - University of California, Berkeley, Berkeley, California
  - Los Angeles County, Los Angeles, California
  - Orange County, Orange, California
  - Clark County, Las Vegas, Nevada
  - Oregon, Bend, Oregon

IPD SHARING:
Plan to Share IPD: Undecided
Because patient and other protected data are involved, we need to consult with our institutional review board and other collaborators concerning which data can be shared.

REFERENCES:
- [Background] Chen KH, Wells JL, Otero MC, Lwi SJ, Haase CM, Levenson RW. Greater Experience of Negative Non-Target Emotions by Patients with Neurodegenerative Diseases Is Related to Lower Emotional Well-Being in Caregivers. Dement Geriatr Cogn Disord. 2017;44(5-6):245-255. doi: 10.1159/000481132. Epub 2017 Dec 8. PMID 29216633
- [Background] Lwi SJ, Ford BQ, Casey JJ, Miller BL, Levenson RW. Poor caregiver mental health predicts mortality of patients with neurodegenerative disease. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):7319-7324. doi: 10.1073/pnas.1701597114. Epub 2017 Jun 27. PMID 28655841
- [Background] Otero MC, Levenson RW. Lower Visual Avoidance in Dementia Patients Is Associated with Greater Psychological Distress in Caregivers. Dement Geriatr Cogn Disord. 2017;43(5-6):247-258. doi: 10.1159/000468146. Epub 2017 Apr 11. PMID 28395276
- [Background] Brown CL, Lwi SJ, Goodkind MS, Rankin KP, Merrilees J, Miller BL, Levenson RW. Empathic Accuracy Deficits in Patients with Neurodegenerative Disease: Association with Caregiver Depression. Am J Geriatr Psychiatry. 2018 Apr;26(4):484-493. doi: 10.1016/j.jagp.2017.10.012. Epub 2017 Dec 27. PMID 29289452
- [Derived] Bullard BM, Brown CL, Scheffer JA, Toledo AB, Levenson RW. Emotion Regulation Strategies and Mental Health in Dementia Caregivers: The Moderating Role of Gender. Dement Geriatr Cogn Disord. 2024;53(3):128-134. doi: 10.1159/000538398. Epub 2024 Apr 22. PMID 38537622

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that outcomes are only assessed regarding caregiver health and well-being. Patients did not provide any information; therefore, all information reported for demographics and measures is only regarding caregivers.
Period: Overall Study
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Started | 41 | 37
Completed | 34 | 30
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Population: Although 78 individuals originally consented to being in the study, 9 individuals dropped out between consenting/enrolling and completing the baseline questionnaire assessing baseline outcome measures; therefore, these baseline numbers only include 69 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | In-Home Technology System | Limited In-Home Technology System | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.38 (12.70) | 65.91 (10.75) | 65.01 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 12 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 0 | 5
  East Asian, South Asian, Southeast Asian, or Indian American | 2 | 1 | 3
  Latino or Hispanic American | 2 | 2 | 4
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Non-Hispanic White or European American | 24 | 26 | 50
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Interview-Short Form
Description: Questionnaire to measure caregiver burden (Zarit, Reever, & Bach-Peterson, 1980). 12 items are rated on 0-4 scale. Range: 0-48. No subscales. Higher scores represent worse outcomes.
Time Frame: 9 months after baseline
Population: 78 individuals enrolled into the study, 9 individuals dropped out before completing the baseline measure, and another 9 dropped out before completing the 9-month assessment for a total 60 individuals for this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 33 | 27
score on a scale | 24.58 (8.09) | 25.59 (8.44)

2. Primary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: Questionnaire to measure depression (Radloff, 1977). 20 items are rated on a 0-3 scale and summed (range = 0-60). There are no subscales. Higher scores represent worse outcomes. The clinical cut-off is usually set at a score of 16.
Time Frame: 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 34 | 30
score on a scale | 19.21 (12.03) | 19.30 (12.37)

3. Primary Outcome: Beck Anxiety Inventory (BAI)
Description: Questionnaire to measure anxiety (Beck, Epstein, Brown, & Steer, 1988). 20 items are rated on a 0-3 scale and summed (range= 0-60). Higher scores indicate worse outcomes. There are no subscales. A score greater than 36 is considered to be clinically significant.
Time Frame: 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 34 | 30
score on a scale | 7.74 (6.82) | 11.20 (8.08)

4. Primary Outcome: Satisfaction With Life Scale
Description: Questionnaire measuring overall life satisfaction and well-being (Diener, Emmons, Larsen, & Griffin, 1985). 5 items scored on a 1-7 scale and summed (Range = 5-35). Lower scores indicate worse outcomes. A score of 20 is considered neutral with higher scores considered increasingly more satisfied and lower scores considered increasingly more dissatisfied.
Time Frame: 9 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | In-Home Technology System | Limited In-Home Technology System
Number analyzed (Participants) | 34 | 30
score on a scale | 17.35 (7.36) | 19.00 (6.14)

ADVERSE EVENTS:
Time Frame: Baseline to 9 months
Description: Although 78 individuals originally enrolled in the study, only 69 individuals completed the baseline assessment. Therefore, the number for those at risk only reflect the 69 individuals for whom we had a baseline assessment.
Arm/Group | In-Home Technology System | Limited In-Home Technology System
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 0/37 | 0/32

LIMITATIONS AND CAVEATS:
The study intended to recruit 80 participants, 78 individuals did complete the consent form, however towards the end of enrollment, COVID-19 shutdowns occurred and our local IRB (UC Berkeley) did not allow in-person contact with participants, which ruled out the ability to install the treatment (technology) in participants' homes. The total number of participants was 69.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03828383/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03828383/SAP_001.pdf